CLINICAL TRIAL: NCT02327000
Title: A Randomized, Open-label, Single Dose, Parallel Study to Evaluate the Pharmacokinetics Dose Proportionality of GLA5PR GLARS-NF1 Tablet in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GL Pharm Tech Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: GLA5PR-104
Record Dates: First submitted 2014-12-10; First posted 2014-12-30 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Healthy
MeSH Terms: interventions — Pregabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- GLA5PR GLARS-NF1 tablet 150mg (Experimental): GLA5PR GLARS-NF1 tablet 150mg/day(Pregabalin 150mg once a day, after meal)
  Interventions: Drug: Pregabalin 150mg
- GLA5PR GLARS-NF1 tablet 300mg (Experimental): GLA5PR GLARS-NF1 tablet 300mg/day(Pregabalin 300mg once a day, after meal)
  Interventions: Drug: Pregabalin 300mg
- GLA5PR GLARS-NF1 tablet 450mg (Experimental): GLA5PR GLARS-NF1 tablet 450mg/day(Pregabalin 150mg 1 tablet and Pregabalin 300mg 1 tablet, 1 times a day, after meal)
  Interventions: Drug: Pregabalin 150mg; Drug: Pregabalin 300mg
- GLA5PR GLARS-NF1 tablet 600mg (Experimental): GLA5PR GLARS-NF1 tablet 600mg/day(Pregabalin 300mg, 2 tablets 1 times a day, after meal)
  Interventions: Drug: Pregabalin 300mg

INTERVENTIONS:
Drug: Pregabalin 150mg — GLA5PR GLARS-NF1 tablet 150mg/day(Pregabalin 150mg once a day)
  Other Names: GLA5PR GLARS-NF1 tablet 150mg
  Arms: GLA5PR GLARS-NF1 tablet 150mg; GLA5PR GLARS-NF1 tablet 450mg
Drug: Pregabalin 300mg — GLA5PR GLARS-NF1 tablet 300mg/day(Pregabalin 300mg once a day)
  Other Names: GLA5PR GLARS-NF1 tablet 300mg
  Arms: GLA5PR GLARS-NF1 tablet 300mg; GLA5PR GLARS-NF1 tablet 450mg; GLA5PR GLARS-NF1 tablet 600mg

SUMMARY:
The purpose of this clinical trial is to compare the pharmacokinetic characteristics of GLA5PR GLARS tablet 150mg and Lyrica Capsule 75mg.

GLA5PR GLARS tablet 150mg is a New Formulation which is made by GL Pharm Tech.

GLARS(Geometrically Long Absorption Regulated System) is New Solution to Sustained Absorption by Extending the Absorption Site.

To overcome the shortcomings of the currently existing sustained release drug delivery technologies the investigators have recently developed a novel drug delivery system to enable a drug to be dissolved irrespective of the surrounding environment and further absorbed up to colon. The investigators coined this "Geometrically Long Absorption Regulated System(GLARS)".

DETAILED DESCRIPTION:
Basically, this system is a triple-layered tablet, comprised of upper and lower layers that swell and draw a sufficient amount of water, plus a highly water - soluble middle layer that rapidly draw water into the tablet core simultaneously.

The water drawn into the tablet (about 3 to 4 times the weight of the tablet itself) functions as an additional media which enables additional and later drug release out of the dosage form. This serves to overcome the shortage of surrounding media that has been reported to be one of the key reasons for mal-absorption of a drug in colon.

As the middle layer induces a rapid water draw into the tablet core, the penetrated water also diffuses to the upper and lower layers, which makes the tablet to rapidly swell and controls drug release.

At virtually the same time, the swollen upper and lower layers form to surround a lateral side of the middle layer, which can, in turn, further control drug release.

This relatively rigid swollen matrix structure makes drug release not affected by surrounding mechanical flux, which can provide relatively consistent in vivo drug release irrespective of degree of gastrointestinal motility.

ELIGIBILITY:
Inclusion Criteria:

* 19~45 years old, Healthy Adult Male Subject
* 17.5~30.5kg/m2(BMI) and ≥ 40kg(Body Weight)

Exclusion Criteria:

* SBP ≥ 140mmHg or DBP ≥ 90mmHg

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-10; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
AUClast | 36hrs
  Pharmacokinetic of Pregabalin
Cmax | 36hrs
  Pharmacokinetic of Pregabalin

SECONDARY OUTCOMES:
AUCinf | 36hrs
  Pharmacokinetic of Pregabalin
Tmax | 36hrs
  Pharmacokinetic of Pregabalin
t1/2 | 36hrs
  Pharmacokinetic of Pregabalin
CL/F | 36hrs
  Pharmacokinetic of Pregabalin
Vd/F | 36hrs
  Pharmacokinetic of Pregabalin

REFERENCES:
- [Derived] Shin KH, Jeon JY, Jang K, Kim TE, Kim MG. Dose-proportional pharmacokinetic properties of GLA5PR GLARS-NF1 controlled-release pregabalin in healthy Korean volunteers: a randomized, open, single-dose, parallel study. Drug Des Devel Ther. 2018 Oct 11;12:3449-3457. doi: 10.2147/DDDT.S167668. eCollection 2018. PMID 30349198